CLINICAL TRIAL: NCT00665925
Title: A Phase II, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Dose Study of Two Doses of R935788 in Rheumatoid Arthritis Patients Failing to Respond to Methotrexate
Brief Title: Efficacy and Safety Study of R935788 Tablets to Treat Rheumatoid Arthritis
Acronym: Taski-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigel Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-935788-010
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Results first posted 2016-06-13 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — fostamatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): R788, 100 mg tablet, orally, twice-a-day
  Interventions: Drug: Fostamatinib disodium (R935788)
- 2 (Experimental): R788, 150 mg tablet, orally, once a day
  Interventions: Drug: Fostamatinib disodium (R935788)
- 3 (Placebo Comparator): Placebo, orally, either once a day, or twice a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fostamatinib disodium (R935788) — 100 mg tablet, orally, twice-a-day
  Other Names: R935788
  Arms: 1
Drug: Fostamatinib disodium (R935788) — 150 mg tablet, orally, once a day
  Other Names: R935788
  Arms: 2
Drug: Placebo — Placebo, orally, either once a day, or twice a day
  Arms: 3

SUMMARY:
The purpose of this study is to determine whether the Spleen Tyrosine Kinase (Syk) inhibitor, R935788 (R788), at a dose of 100 mg, orally, twice-a-day, and/or a dose of of 150 mg, orally, once-a-day is effective in the treatment of Rheumatoid Arthrits in patients who have had an inadequate clinical response to methotrexate.

ELIGIBILITY:
Inclusion Criteria:

* Patients must give written informed consent by signing an IRB/EC-approved Informed Consent Form (ICF) prior to admission to this study.
* Males and females, 18 years of age or older, with active RA for at least 6 months prior to Day 1 dosing.
* Patients must have been receiving weekly methotrexate doses (7.5-25 mg/week) for a minimum of 3 months prior to Day 1 dosing and must be receiving a stable MTX dose, with no change in route, for the previous 6 weeks prior to Day 1 dosing.

'Patients must be receiving a folic or folinic acid supplementation at a stable dose for at least 6 weeks prior to Day 1 dosing.

* Females of childbearing potential must be fully informed of the potential for R788 to adversely affect the fetus and, if sexually active, must agree to use a well established method of birth control during the study (oral contraceptive, mechanical barrier, long acting hormonal agent). These patients must not be lactating and must have a negative urine pregnancy test at the time of randomization and at each laboratory determination.
* The patient must otherwise be in good health as determined by the Investigator on the basis of medical history, physical examination, and laboratory screening tests during the screening period. See exclusion criteria for specific exclusions.
* In the Investigator's opinion, the patient has the ability to understand the nature of the study and any hazards of participation, and to communicate satisfactorily with the Investigator and to participate in, and to comply with, the requirements of the entire protocol.

Exclusion Criteria:

* The patient has a history of, or a concurrent, clinically significant illness, medical condition (other than arthritis) or laboratory abnormality that, in the Investigator's opinion, could affect the conduct of the study. Specifically, excluded are patients with the following:

  1. uncontrolled or poorly controlled hypertension;
  2. other autoimmune disease (psoriatic arthritis, lupus, mixed connective disorder) or arthritis syndromes (gout, Lyme disease, Reiter's syndrome);
  3. recent (within past 2 months prior to Day 1 dosing) serious surgery or infectious disease;
  4. recent history (past 5 years prior to Day 1 dosing) of, or treatment for, a malignancy other than nonmelanomatous skin cancer, or any history of lymphoma;
  5. Hepatitis B ;
  6. Hepatitis C ;
  7. interstitial pneumonitis or active pulmonary infection on chest x-ray;
  8. Tuberculosis (TB): the TB skin test should be negative.
  9. known laboratory abnormalities.
* The patient has a history of substance abuse, drug addiction or alcoholism. Patients may consume up to 4 units of alcohol per week; however, alcohol should be avoided in the 72 hours prior to lab assessments. Patients who cannot reliably comply with this should be excluded. A unit of alcohol is defined as the following: Beer=12 oz or 355 mL; wine = 5 oz or 148 mL; sweet dessert wine=3 oz or 89 mL; 80 proof distilled spirits= 1.5 oz or 44 mL.
* The patient has been treated previously treated with R788 under a different protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 457 (Actual)
Dates: Start 2008-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel B Magilavy, MD, Study Director — Rigel Pharmaceuticals
Locations (65):
- United States (24):
  - Divison of Rheumatology Allergy and Immunology, La Jolla, California
  - Desert Medical Advances, Palm Desert, California
  - Arthritis & Osteoporosis Center, PC, Hamden, Connecticut
  - Cynthia Morgan, Washington D.C., District of Columbia
  - Florida Medical Research Institute, Gainsville, Florida
  - Paddock Park Clinical Research, Ocala, Florida
  - Jeffrey Poiley, MD, Orlando, Florida
  - Lovelace Scientific Resources, Sarasota, Florida
  - Rheumatology Associates, SC, Chicago, Illinois
  - Memorial Medical Group Clinical Research Inst, South Bend, Indiana
  - Center for Arthritis & Osteoporosis, Elizabethtown, Kentucky
  - The Osteoporosis & Clinical Trials Center, Hagerstown, Maryland
  - Fiechtner Research, Inc., Lansing, Michigan
  - Westroads Medical Group, Omaha, Nebraska
  - North Carolina Arthritis & Allergy Care Center, Raleigh, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Health Research of Oklahoma, Oklahoma City, Oklahoma
  - Rheumatology Associates, Erie, Pennsylvania
  - Clinical Research Center of Reading, LLP, West Reading, Pennsylvania
  - Rheumatic Disease Associates, Willow Grove, Pennsylvania
  - Rheumatology Associates, Charleston, South Carolina
  - Austin Rheumatology & Research, Austin, Texas
  - Arthritis Center of South Texas, San Antonio, Texas
  - Arthritis Northwest, PLLC, Spokane, Washington
- Bulgaria (4):
  - MNTranspH "Tsar Boris Treti", Sofia, Gsof
  - MHAT "Kaspela", Plovdiv, PLO
  - MHAT Ruse, Rousse
  - DCC "Sv. Anna" Sofia, Sofia
- Colombia (9):
  - Unidad Medica Torre Plaza, Medellín, Antioquia
  - Centro de Reumatologia y Ortopedia, Barranquilla, Atlántico
  - Reumatologos del Caribe, Barranquilla, Atlántico
  - CIREEM, Bogota, Cundinamarca
  - Fundación Instituto de Reumatología, Bogota, Cundinamarca
  - Riesgo de Fractura S.A, Bogota, Cundinamarca
  - Private Office, Bogotá, Cundinamarca
  - Centro Medico Carlos Ardila Lulle, Bucaramanga, Santander Department
  - SERVIMED, Bucaramanga, Santander Department
- Mexico (11):
  - Christus Muguerza del Parque, Chihuahua City, Chihuahua
  - Arké Estudios Clínicos S.A de C.V, México, D.f.
  - Clínica para el Diagnostico y Tratamiento de, México, D.f.
  - Hospital Ángeles Metropolitano, México, D.f.
  - Hospital General de México, México, D.f.
  - Hospital Aranda de la Parra, León, Guanajuato
  - Instituto Jalisciense de Investigación Clínica, Guadalajara, Jalisco
  - Hospital Civil de Guadalajara "Fray Antonio A, Guadalajara, Jalisco
  - Centro Médico DALINDE, Mexico City, Mexico City
  - Centro de Investigacion Clinical de Morelia, Morelia, Michoacán
  - Hospital Inovamed , Torre Médica, Cuernavaca, Morelos
- Poland (11):
  - NZOZ Centrum Medyczne Artur Racewicz, Bialystok
  - Szpit. Spec.Nr 1, Odz. Reumatol. i Reh., Bytom
  - Wojewodzki Szpital Zespolony Oddzial Reumatol, Elblag
  - Mazowieckie Centrum Badan Klinicznych, Grodzisk Mazowiecki
  - Malopolskie Centrum Medyczne SC, Krakow
  - Krakowskie Centrum Medyczne NZOZ, Krakow
  - NZOZ Reumed, Lublin
  - NZOZ "Nasz Lekarz", Torun
  - Synexus SCM, Wroclaw
  - ASK Klinika Reumatologii i Chor. Wewn., Wroclaw
  - ZOZ w Zyradowie Oddzial Reumatologii, Zyradow
- Romania (6):
  - Spitalul Clinic Judetean de Urgenta Cluj Reum, Cluj-Napoca, Cluj
  - Spitalul Clinic "Sf. Maria" Med Int si Reumat, Bucharest, Sector 1
  - Spitalul Clinic Judetean Sibiu, Sibiu, Sibiu County
  - CMI "Cristei R. Dorica", Brăila
  - Spitalul de Urgenta al MAI Dr. D. Gerota, Bucharest
  - Spitalul Judetean "Dr. Fogolyan Kristol", Sf. Gheorghe

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weinblatt ME, Kavanaugh A, Genovese MC, Musser TK, Grossbard EB, Magilavy DB. An oral spleen tyrosine kinase (Syk) inhibitor for rheumatoid arthritis. N Engl J Med. 2010 Sep 30;363(14):1303-12. doi: 10.1056/NEJMoa1000500. Epub 2010 Sep 22. PMID 20879879

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant received the first dose of study drug on 19 May 2008; the last participant completed the study on 01 June 2009. Participants were recruited from centers in the United States, Europe and Latin America.
Pre-assignment Details: Male/female participants who had active rheumatoid arthritis (RA) for a minimum of 6 months, and receiving a weekly methotrexate (MTX) dose for a minimum of 3 months were randomly assigned to receive R788 150 mg once daily, 100 mg twice daily, placebo once daily or placebo twice daily. It was planned to randomize approximately 420 participants.
Groups:
- Placebo qd: Placebo to R788, oral tablets, once daily, double-blind
- Placebo Bid: Placebo to R788, oral tablets, twice daily, double-blind
- R788 150 mg qd: R788 150 mg, oral tablets, once daily, double-blind
- R788 100 mg Bid: R788 100 mg, oral tablets, twice daily, double-blind
Period: Overall Study
Arm/Group | Placebo qd | Placebo Bid | R788 150 mg qd | R788 100 mg Bid
Started | 77 (Participants randomized) | 76 (Participants randomized) | 152 (Participants randomized) | 152 (Participants randomized)
Completed | 62 (Participants completed the study) | 59 (Participants completed the study) | 126 (Participants completed the study) | 131 (Participants completed the study)
Not Completed | 15 | 17 | 26 | 21
Not completed — Lack of Efficacy | 10 | 8 | 9 | 8
Not completed — Lost to Follow-up | 1 | 2 | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2 | 3 | 2
Not completed — Physician Decision | 0 | 0 | 1 | 2
Not completed — Severe Non-Compliance to Protocol | 0 | 0 | 1 | 1
Not completed — Adverse Event | 1 | 5 | 10 | 5
Not completed — Enrolled by mistake | 0 | 0 | 0 | 1
Not completed — Due to exclusion criteria | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo qd | Placebo Bid | R788 150 mg qd | R788 100 mg Bid | Total
Number analyzed (Participants) | 77 | 76 | 152 | 152 | 457
Age, Continuous [Mean (Standard Deviation); unit: Years] — Please note, baseline data were only calculated for the placebo qd and placebo bid groups. Data from the placebo groups were only pooled for the efficacy analyses.
  Years | 51.3 (13.68) | 53.4 (12.66) | 52.6 (12.31) | 52.5 (12.97) | 52.5 (12.80)
Sex: Female, Male [Count of Participants; unit: Participants] — Please note, baseline data were only calculated for the placebo qd and placebo bid groups. Data from the placebo groups were only pooled for the efficacy analyses.
  Participants
    Female | 67 | 64 | 128 | 131 | 390
    Male | 10 | 12 | 24 | 21 | 67

OUTCOME MEASURES:

1. Primary Outcome: American College of Rheumatology 20 (ACR20) Response at 6 Months
Description: The number of participants with greater than or equal to 20% improvement in tender and swollen joint counts, AND in any 3 of the following: physician's assessment of disease activity, patient's assessment of disease activity, patient's assessment of pain, HAQ-DI; and C-Reactive Protein (CRP) or erythrocyte sedimentation rate (ESR), after 6 months
Time Frame: 6 months
Population: Intent-to-treat population includes all subjects that received study drug
Measure: Number; unit: Participants
Groups:
- Arm 1 - Placebo qd: Placebo to R788, oral tablets, once daily, double-blind
- Arm 2 - Placebo Bid: Placebo to R788, oral tablets, twice daily, double-blind
- Arm 3 - Placebo Pooled: Placebo to R788, oral tablets once and twice daily pooled
- Arm 4 - R788 150 mg qd: R788 150 mg, oral tablets, once daily, double-blind
- Arm 5 - R788 100 mg Bid: R788 100 mg, oral tablets, twice daily, double-blind
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 153 | 152 | 151
Participants |  |  | 53 | 87 | 101

2. Secondary Outcome: American College of Rheumatology 20 (ACR20) Response at 1 Week
Description: The number of participants with greater than or equal to 20% improvement in tender and swollen joint counts, AND in any 3 of the following: physician's assessment of disease activity, patient's assessment of disease activity, patient's assessment of pain, HAQ-DI; and C-Reactive Protein (CRP) or erythrocyte sedimentation rate (ESR), after 1 week
Time Frame: 1 week
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 153 | 151 | 146
Participants |  |  | 21 | 34 | 53

3. Secondary Outcome: American College of Rheumatology 20 (ACR20) Response at 2 Weeks
Description: The number of participants with greater than or equal to 20% improvement in tender and swollen joint counts, AND in any 3 of the following: physician's assessment of disease activity, patient's assessment of disease activity, patient's assessment of pain, HAQ-DI; and C-Reactive Protein (CRP) or erythrocyte sedimentation rate (ESR), after 2 weeks
Time Frame: 2 weeks
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 153 | 152 | 148
Participants |  |  | 29 | 47 | 67

4. Secondary Outcome: American College of Rheumatology 20 (ACR20) Response at 1 Month
Description: The number of participants with greater than or equal to 20% improvement in tender and swollen joint counts, AND in any 3 of the following: physician's assessment of disease activity, patient's assessment of disease activity, patient's assessment of pain, HAQ-DI; and C-Reactive Protein (CRP) or erythrocyte sedimentation rate (ESR), after 1 month
Time Frame: 1 month
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 151 | 152 | 150
Participants |  |  | 48 | 72 | 89

5. Secondary Outcome: American College of Rheumatology 20 (ACR20) Response at 6 Weeks
Description: The number of participants with greater than or equal to 20% improvement in tender and swollen joint counts, AND in any 3 of the following: physician's assessment of disease activity, patient's assessment of disease activity, patient's assessment of pain, HAQ-DI; and C-Reactive Protein (CRP) or erythrocyte sedimentation rate (ESR), after 6 weeks
Time Frame: 6 weeks
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 148 | 151 | 150
Participants |  |  | 55 | 75 | 84

6. Secondary Outcome: American College of Rheumatology 20 (ACR20) Response at 2 Months
Description: The number of participants with greater than or equal to 20% improvement in tender and swollen joint counts, AND in any 3 of the following: physician's assessment of disease activity, patient's assessment of disease activity, patient's assessment of pain, HAQ-DI; and C-Reactive Protein (CRP) or erythrocyte sedimentation rate (ESR), after 2 months
Time Frame: 2 months
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 151 | 151 | 149
Participants |  |  | 58 | 81 | 95

7. Secondary Outcome: American College of Rheumatology 20 (ACR20) Response at 3 Months
Description: The number of participants with greater than or equal to 20% improvement in tender and swollen joint counts, AND in any 3 of the following: physician's assessment of disease activity, patient's assessment of disease activity, patient's assessment of pain, HAQ-DI; and C-Reactive Protein (CRP) or erythrocyte sedimentation rate (ESR), after 3 months
Time Frame: 3 months
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 152 | 152 | 150
Participants |  |  | 64 | 79 | 97

8. Secondary Outcome: American College of Rheumatology 20 (ACR20) Response at 4 Months
Description: The number of participants with greater than or equal to 20% improvement in tender and swollen joint counts, AND in any 3 of the following: physician's assessment of disease activity, patient's assessment of disease activity, patient's assessment of pain, HAQ-DI; and C-Reactive Protein (CRP) or erythrocyte sedimentation rate (ESR), after 4 months
Time Frame: 4 months
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 152 | 151 | 147
Participants |  |  | 57 | 71 | 100

9. Secondary Outcome: American College of Rheumatology 20 (ACR20) Response at 5 Months
Description: The number of participants with greater than or equal to 20% improvement in tender and swollen joint counts, AND in any 3 of the following: physician's assessment of disease activity, patient's assessment of disease activity, patient's assessment of pain, HAQ-DI; and C-Reactive Protein (CRP) or erythrocyte sedimentation rate (ESR), after 5 months
Time Frame: 5 months
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 151 | 152 | 150
Participants |  |  | 61 | 84 | 97

10. Secondary Outcome: American College of Rheumatology 50 (ACR50) Response at 1 Week
Description: The number of participants with greater than or equal to 50% improvement in tender and swollen joint counts, AND in any 3 of the following: physician's assessment of disease activity, patient's assessment of disease activity, patient's assessment of pain, HAQ-DI; and C-Reactive Protein (CRP) or erythrocyte sedimentation rate (ESR), after 1 week
Time Frame: 1 week
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 153 | 151 | 146
Participants |  |  | 4 | 7 | 10

11. Secondary Outcome: American College of Rheumatology 50 (ACR50) Response at 2 Weeks
Description: The number of participants with greater than or equal to 50% improvement in tender and swollen joint counts, AND in any 3 of the following: physician's assessment of disease activity, patient's assessment of disease activity, patient's assessment of pain, HAQ-DI; and C-Reactive Protein (CRP) or erythrocyte sedimentation rate (ESR), after 2 weeks
Time Frame: 2 weeks
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 153 | 152 | 148
Participants |  |  | 7 | 15 | 21

12. Secondary Outcome: American College of Rheumatology 50 (ACR50) Response at 1 Month
Description: The number of participants with greater than or equal to 50% improvement in tender and swollen joint counts, AND in any 3 of the following: physician's assessment of disease activity, patient's assessment of disease activity, patient's assessment of pain, HAQ-DI; and C-Reactive Protein (CRP) or erythrocyte sedimentation rate (ESR), after 1 month
Time Frame: 1 month
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 151 | 152 | 150
Participants |  |  | 11 | 24 | 45

13. Secondary Outcome: American College of Rheumatology 50 (ACR50) Response at 6 Weeks
Description: The number of participants with greater than or equal to 50% improvement in tender and swollen joint counts, AND in any 3 of the following: physician's assessment of disease activity, patient's assessment of disease activity, patient's assessment of pain, HAQ-DI; and C-Reactive Protein (CRP) or erythrocyte sedimentation rate (ESR), after 6 weeks
Time Frame: 6 weeks
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 148 | 151 | 150
Participants |  |  | 19 | 30 | 43

14. Secondary Outcome: American College of Rheumatology 50 (ACR50) Response at 2 Months
Description: The number of participants with greater than or equal to 50% improvement in tender and swollen joint counts, AND in any 3 of the following: physician's assessment of disease activity, patient's assessment of disease activity, patient's assessment of pain, HAQ-DI; and C-Reactive Protein (CRP) or erythrocyte sedimentation rate (ESR), after 2 months
Time Frame: 2 months
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 151 | 151 | 149
Participants |  |  | 22 | 34 | 51

15. Secondary Outcome: American College of Rheumatology 50 (ACR50) Response at 3 Months
Description: The number of participants with greater than or equal to 50% improvement in tender and swollen joint counts, AND in any 3 of the following: physician's assessment of disease activity, patient's assessment of disease activity, patient's assessment of pain, HAQ-DI; and C-Reactive Protein (CRP) or erythrocyte sedimentation rate (ESR), after 3 months
Time Frame: 3 months
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 152 | 152 | 150
Participants |  |  | 23 | 43 | 58

16. Secondary Outcome: American College of Rheumatology 50 (ACR50) Response at 4 Months
Description: The number of participants with greater than or equal to 50% improvement in tender and swollen joint counts, AND in any 3 of the following: physician's assessment of disease activity, patient's assessment of disease activity, patient's assessment of pain, HAQ-DI; and C-Reactive Protein (CRP) or erythrocyte sedimentation rate (ESR), after 4 months
Time Frame: 4 months
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 152 | 151 | 147
Participants |  |  | 25 | 34 | 62

17. Secondary Outcome: American College of Rheumatology 50 (ACR50) Response at 5 Months
Description: The number of participants with greater than or equal to 50% improvement in tender and swollen joint counts, AND in any 3 of the following: physician's assessment of disease activity, patient's assessment of disease activity, patient's assessment of pain, HAQ-DI; and C-Reactive Protein (CRP) or erythrocyte sedimentation rate (ESR), after 5 months
Time Frame: 5 months
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 151 | 152 | 150
Participants |  |  | 25 | 41 | 62

18. Secondary Outcome: American College of Rheumatology 50 (ACR50) Response at 6 Months
Description: The number of participants with greater than or equal to 50% improvement in tender and swollen joint counts, AND in any 3 of the following: physician's assessment of disease activity, patient's assessment of disease activity, patient's assessment of pain, HAQ-DI; and C-Reactive Protein (CRP) or erythrocyte sedimentation rate (ESR), after 6 months
Time Frame: 6 months
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 153 | 152 | 151
Participants |  |  | 29 | 49 | 65

19. Secondary Outcome: American College of Rheumatology 70 (ACR70) Response at 1 Week
Description: The number of participants with greater than or equal to 70% improvement in tender and swollen joint counts, AND in any 3 of the following: physician's assessment of disease activity, patient's assessment of disease activity, patient's assessment of pain, HAQ-DI; and C-Reactive Protein (CRP) or erythrocyte sedimentation rate (ESR), after 1 week
Time Frame: 1 week
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 153 | 151 | 146
Participants |  |  | 1 | 1 | 2

20. Secondary Outcome: American College of Rheumatology 70 (ACR70) Response at 2 Weeks
Description: The number of participants with greater than or equal to 70% improvement in tender and swollen joint counts, AND in any 3 of the following: physician's assessment of disease activity, patient's assessment of disease activity, patient's assessment of pain, HAQ-DI; and C-Reactive Protein (CRP) or erythrocyte sedimentation rate (ESR), after 2 weeks
Time Frame: 2 weeks
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 153 | 152 | 148
Participants |  |  | 1 | 5 | 7

21. Secondary Outcome: American College of Rheumatology 70 (ACR70) Response at 1 Month
Description: The number of participants with greater than or equal to 70% improvement in tender and swollen joint counts, AND in any 3 of the following: physician's assessment of disease activity, patient's assessment of disease activity, patient's assessment of pain, HAQ-DI; and C-Reactive Protein (CRP) or erythrocyte sedimentation rate (ESR), after 1 month
Time Frame: 1 month
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 151 | 152 | 150
Participants |  |  | 7 | 13 | 14

22. Secondary Outcome: American College of Rheumatology 70 (ACR70) Response at 6 Weeks
Description: The number of participants with greater than or equal to 70% improvement in tender and swollen joint counts, AND in any 3 of the following: physician's assessment of disease activity, patient's assessment of disease activity, patient's assessment of pain, HAQ-DI; and C-Reactive Protein (CRP) or erythrocyte sedimentation rate (ESR), after 6 weeks
Time Frame: 6 weeks
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 148 | 151 | 150
Participants |  |  | 5 | 13 | 16

23. Secondary Outcome: American College of Rheumatology 70 (ACR70) Response at 2 Months
Description: The number of participants with greater than or equal to 70% improvement in tender and swollen joint counts, AND in any 3 of the following: physician's assessment of disease activity, patient's assessment of disease activity, patient's assessment of pain, HAQ-DI; and C-Reactive Protein (CRP) or erythrocyte sedimentation rate (ESR), after 2 months
Time Frame: 2 months
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 151 | 151 | 149
Participants |  |  | 4 | 15 | 20

24. Secondary Outcome: American College of Rheumatology 70 (ACR70) Response at 3 Months
Description: The number of participants with greater than or equal to 70% improvement in tender and swollen joint counts, AND in any 3 of the following: physician's assessment of disease activity, patient's assessment of disease activity, patient's assessment of pain, HAQ-DI; and C-Reactive Protein (CRP) or erythrocyte sedimentation rate (ESR), after 3 months
Time Frame: 3 months
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 152 | 152 | 150
Participants |  |  | 10 | 19 | 30

25. Secondary Outcome: American College of Rheumatology 70 (ACR70) Response at 4 Months
Description: The number of participants with greater than or equal to 70% improvement in tender and swollen joint counts, AND in any 3 of the following: physician's assessment of disease activity, patient's assessment of disease activity, patient's assessment of pain, HAQ-DI; and C-Reactive Protein (CRP) or erythrocyte sedimentation rate (ESR), after 4 months
Time Frame: 4 months
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 152 | 151 | 147
Participants |  |  | 8 | 17 | 32

26. Secondary Outcome: American College of Rheumatology 70 (ACR70) Response at 5 Months
Description: The number of participants with greater than or equal to 70% improvement in tender and swollen joint counts, AND in any 3 of the following: physician's assessment of disease activity, patient's assessment of disease activity, patient's assessment of pain, HAQ-DI; and C-Reactive Protein (CRP) or erythrocyte sedimentation rate (ESR), after 5 months
Time Frame: 5 months
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 151 | 152 | 150
Participants |  |  | 8 | 20 | 33

27. Secondary Outcome: American College of Rheumatology 70 (ACR70) Response at 6 Months
Description: The number of participants with greater than or equal to 70% improvement in tender and swollen joint counts, AND in any 3 of the following: physician's assessment of disease activity, patient's assessment of disease activity, patient's assessment of pain, HAQ-DI; and C-Reactive Protein (CRP) or erythrocyte sedimentation rate (ESR), after 6 months
Time Frame: 6 months
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 153 | 152 | 151
Participants |  |  | 16 | 21 | 43

28. Secondary Outcome: American College of Rheumatology Index of Improvement (ACRn) at 1 Week
Description: The index of improvement in RA, where 0 indicates no improvement and 100 indicates a 100% improvement across all signs and symptoms of RA after 1 week of treatment
Time Frame: 1 week
Population: Intent-to-treat population with available data and received study drug.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 153 | 151 | 145
Score |  |  | 7.07 (13.677) | 10.75 (15.788) | 16.22 (19.564)

29. Secondary Outcome: American College of Rheumatology Index of Improvement (ACRn) at 2 Weeks
Description: The index of improvement in RA, where 0 indicates no improvement and 100 indicates a 100% improvement across all signs and symptoms of RA after 2 weeks of treatment
Time Frame: 2 weeks
Population: Intent-to-treat population with available data and received study drug.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 151 | 150 | 145
Score |  |  | 9.74 (16.987) | 16.27 (20.899) | 21.62 (23.491)

30. Secondary Outcome: American College of Rheumatology Index of Improvement (ACRn) at 1 Month
Description: The index of improvement in RA, where 0 indicates no improvement and 100 indicates a 100% improvement across all signs and symptoms of RA after 1 month of treatment
Time Frame: 1 month
Population: Intent-to-treat population with available data and received study drug.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 149 | 148 | 146
Score |  |  | 14.65 (20.537) | 24.14 (25.428) | 32.23 (26.304)

31. Secondary Outcome: American College of Rheumatology Index of Improvement (ACRn) at 6 Weeks
Description: The index of improvement in RA, where 0 indicates no improvement and 100 indicates a 100% improvement across all signs and symptoms of RA after 6 weeks of treatment
Time Frame: 6 weeks
Population: Intent-to-treat population with available data and received study drug.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 145 | 146 | 146
Score |  |  | 18.05 (22.904) | 26.87 (26.893) | 31.08 (27.789)

32. Secondary Outcome: American College of Rheumatology Index of Improvement (ACRn) at 2 Months
Description: The index of improvement in RA, where 0 indicates no improvement and 100 indicates a 100% improvement across all signs and symptoms of RA after 2 months of treatment
Time Frame: 2 months
Population: Intent-to-treat population with available data and received study drug.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 148 | 145 | 143
Score |  |  | 20.12 (23.179) | 29.11 (26.827) | 36.73 (28.254)

33. Secondary Outcome: American College of Rheumatology Index of Improvement (ACRn) at 3 Months
Description: The index of improvement in RA, where 0 indicates no improvement and 100 indicates a 100% improvement across all signs and symptoms of RA after 3 months of treatment
Time Frame: 3 months
Population: Intent-to-treat population with available data and received study drug.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 147 | 141 | 142
Score |  |  | 22.11 (25.904) | 31.79 (27.959) | 39.04 (30.059)

34. Secondary Outcome: American College of Rheumatology Index of Improvement (ACRn) at 4 Months
Description: The index of improvement in RA, where 0 indicates no improvement and 100 indicates a 100% improvement across all signs and symptoms of RA after 4 months of treatment
Time Frame: 4 months
Population: Intent-to-treat population with available data and received study drug.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 130 | 130 | 132
Score |  |  | 22.61 (25.661) | 30.24 (28.347) | 44.70 (29.729)

35. Secondary Outcome: American College of Rheumatology Index of Improvement (ACRn) at 5 Months
Description: The index of improvement in RA, where 0 indicates no improvement and 100 indicates a 100% improvement across all signs and symptoms of RA after 5 months of treatment
Time Frame: 5 months
Population: Intent-to-treat population with available data and received study drug.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 123 | 126 | 130
Score |  |  | 25.66 (25.734) | 35.35 (27.683) | 44.76 (29.972)

36. Secondary Outcome: American College of Rheumatology Index of Improvement (ACRn) at 6 Months
Description: The index of improvement in RA, where 0 indicates no improvement and 100 indicates a 100% improvement across all signs and symptoms of RA after 6 months of treatment
Time Frame: 6 months
Population: Intent-to-treat population with available data and received study drug.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 121 | 126 | 130
Score |  |  | 26.00 (29.402) | 38.45 (29.108) | 49.55 (30.189)

37. Secondary Outcome: Disease Activity Score-C-Reactive Protein (DAS28-CRP) <2.6 at 1 Month
Description: Number of participants with DAS28-CRP (measuring RA symptoms including: tender joint count, swollen joint count, patient's assessment of disease activity, and CRP in patients with high CRP at baseline), of less than 2.6. The DAS runs from 0 to 10 - higher scores indicate worse symptoms. A score of less than 2.6 indicates remission of RA symptoms
Time Frame: 1 month
Population: Intent-to-Treat Population with CRP as Primary Phase Reactant with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 85 | 93 | 86
Participants |  |  | 2 | 10 | 4

38. Secondary Outcome: Disease Activity Score-C-Reactive Protein (DAS28-CRP) <2.6 at 2 Months
Description: as for outcome 37
Time Frame: 2 months
Population: Intent-to-Treat Population with CRP as Primary Phase Reactant with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 83 | 94 | 82
Participants |  |  | 3 | 8 | 8

39. Secondary Outcome: Disease Activity Score-C-Reactive Protein (DAS28-CRP) <2.6 at 3 Months
Description: as for outcome 37
Time Frame: 3 months
Population: Intent-to-Treat Population with CRP as Primary Phase Reactant with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 83 | 92 | 84
Participants |  |  | 5 | 7 | 11

40. Secondary Outcome: Disease Activity Score-C-Reactive Protein (DAS28-CRP) <2.6 at 4 Months
Description: as for outcome 37
Time Frame: 4 months
Population: Intent-to-Treat Population with CRP as Primary Phase Reactant with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 73 | 84 | 80
Participants |  |  | 4 | 10 | 15

41. Secondary Outcome: Disease Activity Score-C-Reactive Protein (DAS28-CRP) <2.6 at 5 Months
Description: as for outcome 37
Time Frame: 5 months
Population: Intent-to-Treat Population with CRP as Primary Phase Reactant with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 71 | 81 | 76
Participants |  |  | 5 | 8 | 24

42. Secondary Outcome: Disease Activity Score-C-Reactive Protein (DAS28-CRP) <2.6 at 6 Months
Description: as for outcome 37
Time Frame: 6 months
Population: Intent-to-Treat Population with CRP as Primary Phase Reactant with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 70 | 81 | 77
Participants |  |  | 6 | 17 | 20

43. Secondary Outcome: Disease Activity Score-C-Reactive Protein (DAS28-CRP) <3.2 at 1 Month
Description: Number of participants with DAS28-CRP (measuring RA symptoms including: tender joint count, swollen joint count, patient's assessment of disease activity, and CRP in patients with high CRP at baseline), of less than 3.2. The DAS runs from 0 to 10 - higher scores indicate worse symptoms. A score of less than 3.2 indicates low disease activity
Time Frame: 1 month
Population: Intent-to-Treat Population with CRP as Primary Phase Reactant with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 85 | 93 | 86
Participants |  |  | 6 | 15 | 15

44. Secondary Outcome: Disease Activity Score-C-Reactive Protein (DAS28-CRP) <3.2 at 2 Months
Description: as for outcome 43
Time Frame: 2 months
Population: Intent-to-Treat Population with CRP as Primary Phase Reactant with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 83 | 94 | 82
Participants |  |  | 9 | 19 | 21

45. Secondary Outcome: Disease Activity Score-C-Reactive Protein (DAS28-CRP) <3.2 at 3 Months
Description: as for outcome 43
Time Frame: 3 months
Population: Intent-to-Treat Population with CRP as Primary Phase Reactant with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 83 | 92 | 84
Participants |  |  | 8 | 25 | 21

46. Secondary Outcome: Disease Activity Score-C-Reactive Protein (DAS28-CRP) <3.2 at 4 Months
Description: as for outcome 43
Time Frame: 4 months
Population: Intent-to-Treat Population with CRP as Primary Phase Reactant with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 73 | 84 | 80
Participants |  |  | 9 | 20 | 28

47. Secondary Outcome: Disease Activity Score-C-Reactive Protein (DAS28-CRP) <3.2 at 5 Months
Description: as for outcome 43
Time Frame: 5 months
Population: Intent-to-Treat Population with CRP as Primary Phase Reactant with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 71 | 81 | 76
Participants |  |  | 8 | 21 | 34

48. Secondary Outcome: Disease Activity Score-C-Reactive Protein (DAS28-CRP) <3.2 at 6 Months
Description: as for outcome 43
Time Frame: 6 months
Population: Intent-to-Treat Population with CRP as Primary Phase Reactant with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 70 | 81 | 77
Participants |  |  | 7 | 26 | 30

49. Secondary Outcome: Disease Activity Score-Erythrocyte Sedimentation Rate (DAS28-ESR) <2.6 at 1 Month
Description: Number of participants with DAS28-ESR (measuring RA symptoms including: tender joint count, swollen joint count, patient's assessment of disease activity, and ESR in patients with high ESR at baseline), of less than 2.6. The DAS runs from 0 to 10 - higher scores indicate worse symptoms. A score of less than 2.6 indicates remission of RA symptoms
Time Frame: 1 month
Population: Intent-to-Treat Population with ESR as Primary Phase Reactant with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 64 | 53 | 61
Participants |  |  | 2 | 3 | 12

50. Secondary Outcome: Disease Activity Score-Erythrocyte Sedimentation Rate (DAS28-ESR) <2.6 at 2 Months
Description: as for outcome 49
Time Frame: 2 months
Population: Intent-to-Treat Population with ESR as Primary Phase Reactant with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 64 | 50 | 60
Participants |  |  | 4 | 4 | 13

51. Secondary Outcome: Disease Activity Score-Erythrocyte Sedimentation Rate (DAS28-ESR) <2.6 at 3 Months
Description: as for outcome 49
Time Frame: 3 months
Population: Intent-to-Treat Population with ESR as Primary Phase Reactant with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 64 | 49 | 58
Participants |  |  | 4 | 3 | 19

52. Secondary Outcome: Disease Activity Score-Erythrocyte Sedimentation Rate (DAS28-ESR) <2.6 at 4 Months
Description: as for outcome 49
Time Frame: 4 months
Population: Intent-to-Treat Population with ESR as Primary Phase Reactant with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 57 | 46 | 53
Participants |  |  | 5 | 3 | 15

53. Secondary Outcome: Disease Activity Score-Erythrocyte Sedimentation Rate (DAS28-ESR) <2.6 at 5 Months
Description: as for outcome 49
Time Frame: 5 months
Population: Intent-to-Treat Population with ESR as Primary Phase Reactant with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 52 | 45 | 54
Participants |  |  | 3 | 7 | 12

54. Secondary Outcome: Disease Activity Score-Erythrocyte Sedimentation Rate (DAS28-ESR) <2.6 at 6 Months
Description: as for outcome 49
Time Frame: 6 months
Population: Intent-to-Treat Population with ESR as Primary Phase Reactant with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 51 | 44 | 54
Participants |  |  | 3 | 9 | 21

55. Secondary Outcome: Disease Activity Score-Erythrocyte Sedimentation Rate (DAS28-ESR) <3.2 at 1 Month
Description: Number of participants with DAS28-ESR (measuring RA symptoms including: tender joint count, swollen joint count, patient's assessment of disease activity, and ESR in patients with high ESR at baseline), of less than 3.2. The DAS runs from 0 to 10 - higher scores indicate worse symptoms. A score of less than 3.2 indicates low disease activity
Time Frame: 1 month
Population: Intent-to-Treat Population with ESR as Primary Phase Reactant with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 64 | 53 | 61
Participants |  |  | 3 | 6 | 18

56. Secondary Outcome: Disease Activity Score-Erythrocyte Sedimentation Rate (DAS28-ESR) <3.2 at 2 Months
Description: as for outcome 55
Time Frame: 2 months
Population: Intent-to-Treat Population with ESR as Primary Phase Reactant with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 64 | 50 | 60
Participants |  |  | 9 | 7 | 23

57. Secondary Outcome: Disease Activity Score-Erythrocyte Sedimentation Rate (DAS28-ESR) <3.2 at 3 Months
Description: as for outcome 55
Time Frame: 3 months
Population: Intent-to-Treat Population with ESR as Primary Phase Reactant with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 64 | 49 | 58
Participants |  |  | 7 | 8 | 22

58. Secondary Outcome: Disease Activity Score-Erythrocyte Sedimentation Rate (DAS28-ESR) <3.2 at 4 Months
Description: as for outcome 55
Time Frame: 4 months
Population: Intent-to-Treat Population with ESR as Primary Phase Reactant with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 57 | 46 | 53
Participants |  |  | 8 | 6 | 23

59. Secondary Outcome: Disease Activity Score-Erythrocyte Sedimentation Rate (DAS28-ESR) <3.2 at 5 Months
Description: as for outcome 55
Time Frame: 5 months
Population: Intent-to-Treat Population with ESR as Primary Phase Reactant with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 52 | 45 | 54
Participants |  |  | 7 | 8 | 24

60. Secondary Outcome: Disease Activity Score-Erythrocyte Sedimentation Rate (DAS28-ESR) <3.2 at 6 Months
Description: as for outcome 55
Time Frame: 6 months
Population: Intent-to-Treat Population with ESR as Primary Phase Reactant with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 51 | 44 | 54
Participants |  |  | 8 | 11 | 29

61. Secondary Outcome: Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) at 6 Months
Description: Change from baseline in FACIT-F, which is a patient-reported 13-item questionnaire that assesses fatigue, calculated as the score at 6 months minus the score at baseline. The FACIT-F runs from 0 to 52 with lower scores indicating higher fatigue. A positive change from baseline indicates an improvement in fatigue after treatment.
Time Frame: Baseline to 6 months
Population: Intent-to-treat population with available data and received study drug.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 109 | 107 | 117
Score |  |  | 4.5 (9.79) | 5.7 (10.28) | 7.4 (10.87)

62. Secondary Outcome: Short Form Health Survey (SF-36) Physical Component Summary (PCS) at 6 Months
Description: Change from baseline in the PCS of the SF-36 (which assesses health and wellbeing), calculated as the score at 6 months minus the score at baseline. The PCS ranges from 0 to 100 with 100 indicating the highest level of functioning possible. A positive change indicates an improvement in PCS after treatment
Time Frame: Baseline to 6 months
Population: Intent-to-treat population with available data and received study drug.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 118 | 124 | 129
Score |  |  | 4.902 (8.4808) | 5.903 (8.9541) | 8.524 (8.7068)

63. Secondary Outcome: Short Form Health Survey (SF-36) Mental Component Summary (MCS) at 6 Months
Description: Change from baseline in the MCS of the SF-36 (which assesses health and wellbeing), calculated as the score at 6 months minus the score at baseline. The MCS ranges from 0 to 100 with 100 indicating the highest level of functioning possible. A positive change indicates an improvement in MCS after treatment
Time Frame: Baseline to 6 months
Population: Intent-to-treat population with available data and received study drug.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 0 | 0 | 118 | 125 | 129
Score |  |  | 3.711 (10.7098) | 2.033 (10.7089) | 3.990 (10.5129)

64. Secondary Outcome: Alanine Aminotransferase (ALT) >1.5x Upper Limit of Normal (ULN)
Description: The number of participants with ALT (a test of liver function) values greater than 1.5 times the ULN
Time Frame: Any time between baseline and 6 months
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 77 | 76 | 0 | 152 | 152
Participants | 3 | 11 |  | 28 | 31

65. Secondary Outcome: Alanine Aminotransferase (ALT) >1.5-2x Upper Limit of Normal (ULN)
Description: The number of participants with ALT (a test of liver function) values greater than 1.5 to 2 times the ULN
Time Frame: Any time between baseline and 6 months
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 77 | 76 | 0 | 152 | 152
Participants | 1 | 5 |  | 14 | 15

66. Secondary Outcome: Alanine Aminotransferase (ALT) >2-3x Upper Limit of Normal (ULN)
Description: The number of participants with ALT (a test of liver function) values greater than 2 to 3 times the ULN
Time Frame: Any time between baseline and 6 months
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 77 | 76 | 0 | 152 | 152
Participants | 1 | 4 |  | 8 | 10

67. Secondary Outcome: Alanine Aminotransferase (ALT) >3x Upper Limit of Normal (ULN)
Description: The number of participants with ALT (a test of liver function) values greater than 3 times the ULN
Time Frame: Any time between baseline and 6 months
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 77 | 76 | 0 | 152 | 152
Participants | 1 | 2 |  | 6 | 6

68. Secondary Outcome: Alanine Aminotransferase (ALT) >3-5x Upper Limit of Normal (ULN)
Description: The number of participants with ALT (a test of liver function) values greater than 3 to 5 times the ULN
Time Frame: Any time between baseline and 6 months
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 77 | 76 | 0 | 152 | 152
Participants | 1 | 1 |  | 3 | 3

69. Secondary Outcome: Alanine Aminotransferase (ALT) >5-10x Upper Limit of Normal (ULN)
Description: The number of participants with ALT (a test of liver function) values greater than 5 to 10 times the ULN
Time Frame: Any time between baseline and 6 months
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 77 | 76 | 0 | 152 | 152
Participants | 0 | 1 |  | 3 | 3

70. Secondary Outcome: Alanine Aminotransferase (ALT) >10x Upper Limit of Normal (ULN)
Description: The number of participants with ALT (a test of liver function) values greater than 10 times the ULN
Time Frame: Any time between baseline and 6 months
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 77 | 76 | 0 | 152 | 152
Participants | 0 | 0 |  | 0 | 0

71. Secondary Outcome: Aspartate Aminotransferase (AST) >1.5x Upper Limit of Normal (ULN)
Description: The number of participants with AST (a test of liver function) values greater than 1.5 times the ULN
Time Frame: Any time between baseline and 6 months
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 77 | 76 | 0 | 152 | 152
Participants | 1 | 4 |  | 19 | 11

72. Secondary Outcome: Aspartate Aminotransferase (AST) >1.5-2x Upper Limit of Normal (ULN)
Description: The number of participants with AST (a test of liver function) values greater than 1.5-2 times the ULN
Time Frame: Any time between baseline and 6 months
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 77 | 76 | 0 | 152 | 152
Participants | 0 | 1 |  | 13 | 5

73. Secondary Outcome: Aspartate Aminotransferase (AST) >2-3x Upper Limit of Normal (ULN)
Description: The number of participants with AST (a test of liver function) values greater than 2 to 3 times the ULN
Time Frame: Any time between baseline and 6 months
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 77 | 76 | 0 | 152 | 152
Participants | 0 | 2 |  | 4 | 1

74. Secondary Outcome: Aspartate Aminotransferase (AST) >3x Upper Limit of Normal (ULN)
Description: The number of participants with AST (a test of liver function) values greater than 3 times the ULN
Time Frame: Any time between baseline and 6 months
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 77 | 76 | 0 | 152 | 152
Participants | 1 | 1 |  | 2 | 5

75. Secondary Outcome: Aspartate Aminotransferase (AST) >3-5x Upper Limit of Normal (ULN)
Description: The number of participants with AST (a test of liver function) values greater than 3 to 5 times the ULN
Time Frame: Any time between baseline and 6 months
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 77 | 76 | 0 | 152 | 152
Participants | 0 | 1 |  | 2 | 5

76. Secondary Outcome: Aspartate Aminotransferase (AST) >5-10 x Upper Limit of Normal (ULN)
Description: The number of participants with AST (a test of liver function) values greater than 5 to 10 times the ULN
Time Frame: Any time between baseline and 6 months
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 77 | 76 | 0 | 152 | 152
Participants | 1 | 0 |  | 0 | 0

77. Secondary Outcome: Aspartate Aminotransferase (AST) >10 x Upper Limit of Normal (ULN)
Description: The number of participants with AST (a test of liver function) values greater than 10 times the ULN
Time Frame: Any time between baseline and 6 months
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 77 | 76 | 0 | 152 | 152
Participants | 0 | 0 |  | 0 | 0

78. Secondary Outcome: Alkaline Phosphatase >1.5 x Upper Limit of Normal (ULN) and >1.5 Times Baseline
Description: The number of participants with alkaline phosphatase (a test of liver function) values greater than 1.5 times the ULN and greater than 1.5 times baseline
Time Frame: Any time between baseline and 6 months
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 77 | 76 | 0 | 152 | 152
Participants | 0 | 1 |  | 1 | 6

79. Secondary Outcome: Bilirubin >1.5 x Upper Limit of Normal (ULN)
Description: The number of participants with bilirubin (a test of liver function) values greater than 1.5 times the ULN
Time Frame: Any time between baseline and 6 months
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 77 | 76 | 0 | 152 | 152
Participants | 0 | 2 |  | 4 | 4

80. Secondary Outcome: Bilirubin >2 x Upper Limit of Normal (ULN)
Description: The number of participants with bilirubin (a test of liver function) values greater than 2 times the ULN
Time Frame: Any time between baseline and 6 months
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 77 | 76 | 0 | 152 | 152
Participants | 0 | 0 |  | 0 | 3

81. Secondary Outcome: Absolute Neutrophil Count (ANC) <1500/mm3
Description: The number of participants with ANC (a test of liver function) values lower than 1500/mm3
Time Frame: Any time between baseline and 6 months
Population: Intent-to-treat population with available data and received study drug.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo qd | Arm 2 - Placebo Bid | Arm 3 - Placebo Pooled | Arm 4 - R788 150 mg qd | Arm 5 - R788 100 mg Bid
Number analyzed (Participants) | 77 | 76 | 0 | 152 | 152
Participants | 1 | 0 |  | 10 | 9

ADVERSE EVENTS:
Description: Please note, safety data were only calculated for the placebo qd and placebo bid groups. Data from the placebo groups were only pooled for the efficacy analyses
Arm/Group | Placebo qd | Placebo Bid | R788 150 mg qd | R788 100 mg Bid
Serious Adverse Events (participants affected / at risk) | 2/77 | 4/76 | 5/152 | 1/152
Other Adverse Events (participants affected / at risk) | 26/77 | 20/76 | 62/152 | 73/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo qd (N=77) | Placebo Bid (N=76) | R788 150 mg qd (N=152) | R788 100 mg Bid (N=152)
ANGINA UNSTABLE (Cardiac disorders) | 1 | 0 | 1 | 0
DUODENAL ULCER (Gastrointestinal disorders) | 0 | 0 | 0 | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 1
PANCREATITIS (Gastrointestinal disorders) | 0 | 0 | 1 | 0
VOMITING (Gastrointestinal disorders) | 0 | 0 | 0 | 1
ARTHRITIS INFECTIVE (Infections and infestations) | 0 | 1 | 0 | 0
BURSITIS INFECTIVE (Infections and infestations) | 1 | 0 | 0 | 0
CELLULITIS (Infections and infestations) | 0 | 1 | 0 | 1
ERYSIPELAS (Infections and infestations) | 0 | 0 | 1 | 0
GALLBLADDER EMPYEMA (Infections and infestations) | 0 | 0 | 0 | 1
HERPES ZOSTER OPHTHALMIC (Infections and infestations) | 0 | 0 | 0 | 1
OSTEOMYELITIS (Infections and infestations) | 0 | 0 | 0 | 1
PYELONEPHRITIS (Infections and infestations) | 0 | 0 | 1 | 0
SOFT TISSUE INFECTION (Infections and infestations) | 0 | 1 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 1
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
CARCINOMA IN SITU OF PENIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
RENAL CELL CARCINOMA STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 1 | 0 | 0
STILLBIRTH (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
HYDRONEPHROSIS (Renal and urinary disorders) | 0 | 0 | 1 | 0
ASTHMATIC CRISIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo qd (N=77) | Placebo Bid (N=76) | R788 150 mg qd (N=152) | R788 100 mg Bid (N=152)
DIARRHOEA (Gastrointestinal disorders) | 4 | 1 | 18 | 29
NAUSEA (Gastrointestinal disorders) | 1 | 6 | 9 | 7
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 | 2 | 3 | 10
URINARY TRACT INFECTION (Infections and infestations) | 2 | 5 | 5 | 9
INFLUENZA (Infections and infestations) | 2 | 4 | 3 | 5
TRANSAMINASES INCREASED (Investigations) | 3 | 2 | 7 | 8
DYSLIPIDAEMIA (Metabolism and nutrition disorders) | 3 | 2 | 8 | 5
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 | 1 | 1 | 1
HEADACHE (Nervous system disorders) | 3 | 5 | 10 | 9
RASH (Skin and subcutaneous tissue disorders) | 5 | 0 | 2 | 3
HYPERTENSION (Vascular disorders) | 4 | 3 | 18 | 21

LIMITATIONS AND CAVEATS:
The 2 placebo groups (bid and qd) were pooled for all efficacy data summaries and analysis since the observed ACR20 response rate difference between the placebo groups was <15 percentage points (prospectively defined in protocol).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less